CLINICAL TRIAL: NCT06807684
Title: Discerning the Abnormal Functional Connectivity Involving the Social Reciprocity Network in Autism Spectrum Disorder and the Impact of Transcranial Magnetic Stimulation in Mitigating the Abnormalities
Brief Title: Abnormal Connectivity Involving the Social Reciprocity Network in Autism and the Impact of Neurostimulation in Mitigating the Abnormalities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Principal Investigator, Mitra Assadi, Director, Professor of Neurology, Christiana Care Health Services
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DDD 605632
Record Dates: First submitted 2024-08-12; First posted 2025-02-04 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism spectrum; transcranial magnetic stimulation; neuronal connectivity
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: The investigators will recruit ASD cases 13-18 years of age and implementing 18 sessions (3 times/week for 6 weeks) of rTMS or sham stimulation of the bilateral IPL/IFG in a prospective, single blind study design. During phase I (3 weeks), half of the subjects will receive rTMS, while the other half will receive sham stimulation. During phase II (3 weeks) all subjects will receive active stimulation. The investigators will deliver a type of high frequency rTMS known as intermittent theta burst stimulation (iTBS), 2400 stimulations per session, equally divided between the bilateral IPL and IFG.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- phase 1 (Sham Comparator): During phase I (3 weeks), half of the subjects will receive rTMS, while the other half will receive sham stimulation.
  Interventions: Device: transcranial magnetic stimulation
- phase 2 (Active Comparator): During phase II (3 weeks) all subjects will receive active stimulation.
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — The investigators will deliver a type of high frequency rTMS known as intermittent theta burst stimulation (iTBS), 2400 stimulations per session, equally divided between the bilateral IPL and IFG.

SUMMARY:
There is no consensus regarding the neurological substrate underpinning ASD. The investigators describe the novel concept of "social reciprocity network" and hypothesize that aberrant connectivity/oscillatory patterns affecting this network contribute to the core deficits in ASD.

The overarching goal of this trial is to explore abnormalities involving the neuronal connectivity and oscillatory patterns within the social reciprocity network and to elucidate the role of modulating this network via rTMS in improving the above measures and social cognition in ASD. Quantitative electroencephalography (QEEG) coherence and spectral power analysis are reliable measures of neuronal connectivity and dynamics. The investigators aim to study the QEEG coherence/spectral power analysis to explore the neuronal dynamics affecting the social reciprocity network in ASD.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) encompasses a range of limitations in reciprocal and communicative milestones, leading to significant functional challenges throughout the lifespan. While there is no consensus regarding the neuroanatomical substrate underpinning ASD, there are two major schools of thought: a group of researchers have focused on abnormalities affecting the mirror neurons and other cortical areas involved in social reciprocity, while others have proposed a more widespread alteration in neuronal organization in this condition resulting in abnormal white matter trajectories leading to cortical over or under connectivity. The investigators describe the social reciprocity network: the mirror neurons populated in the inferior frontal gyrus (IFG) and inferior parietal lobule (IPL), plus cortical areas involved in abstract social cognition including the medial prefrontal cortex, temporal-parietal junction and posterior cingulate gyrus. We hypothesize that aberrant connectivity affecting the above neuronal circuitry, "the social reciprocity network" contributes significantly to the core deficits in this condition.

Quantitative electroencephalography (QEEG) coherence and spectral power analysis are reliable measures of functional connectivity and neuronal dynamics. The investigators aim to study the QEEG coherence/spectral power analysis to explore the abnormal neuronal dynamics affecting the social reciprocity network in ASD. The existing literature suggest that noninvasive brain modulation, via Repetitive transcranial magnetic stimulation (rTMS), could potentially ameliorate the aberrant connectivity and the behaviors in ASD by altering neuronal dynamics. The investigator's overarching goal is to explore the neuronal connectivity in the social reciprocity network and to elucidate the mechanism of modulating these connections in improving social cognition in ASD.

Within this design, there are 3 aims:

Aim 1: Exploring the QEEG measures of connectivity and oscillatory patterns in the social reciprocity network in ASD. Hypothesis: abnormal connectivity affecting the social reciprocity network contributes to the core deficits in ASD.

Aim 2: Assessing the effects of rTMS of the bilateral social reciprocity network on the connectivity/spectral analysis as well as social cognition in ASD. Hypothesis: neurostimulation of the social reciprocity network ameliorates social cognition, power densities and the functional connectivity within the network.

ELIGIBILITY:
Inclusion criteria

1. Fulfilling the DSM-V criteria for ASD and confirmed by CARS2, HF Exclusion criteria

1. Patients with ASD exhibiting significant anxiety or contact avoidance, precluding them from cooperating with the procedure
2. Patients with a known diagnosis of seizures
3. Presence of any metallic implants or devices in the head or neck area
4. Pregnant women

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Exploring neuronal connectivity and oscillatory patterns in the social reciprocity network in ASD | 9 weeks
  Abnormal connectivity affecting the social reciprocity network contributes to the core deficits in ASD. The investigators will record an electroencephalogram (EEG) at baseline and after completing treatments with transcranial magnetic stimulation. The EEG data will be subjected to mathematical analysis in order to calculate measures of EEG coherence, functional connectivity and oscillatory patterns within the social reciprocity network. These numerical values will be used to discern:
  1. presence of a consistent pattern across the social reciprocity network at baseline for measurements of neuronal connectivity as well as the oscillatory patterns including alpha, beta, gamma, theta and mu rhythms
  2. improvement of the above neuronal connectivity and oscillatory patterns after the transcranial magnetic intervention

SECONDARY OUTCOMES:
Assessing the effects of iTBS stimulation of the bilateral social reciprocity network on social cognition in ASD | 9 weeks
  Presence and severity of autism spectrum disorder as assessed using the Childhood Autism Rating Scale, 2nd addition, high functioning.
  The investigators hypothesize that iTBS of the social reciprocity network ameliorates social cognition in ASD. To measure the outcomes, the investigators will implement the Childhood Autism Rating Scale, 2nd addition, high functioning (CARS2, HF). This is a validated test that is based on actual measures of patient performance on behavioral tasks (score 30-37). The test is administered by a board-certified neuropsychologist before and after neurostimulation intervention. The test produces numerical values quantifying social cognition, reciprocity and rigid behaviors, comparing the results before and after the treatment to discern any potential efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Christiana Care, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
we will enter all the data to the NIMH repository
Supporting Information: Study Protocol, CSR
Time Frame: January thru Dec 2025